CLINICAL TRIAL: NCT02284451
Title: Facilitating HIV/AIDS and HIV Testing Literacy for Emergency Department Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other); Northeastern University (Other); Olive View-UCLA Education & Research Institute (Other); University of Alabama at Birmingham (Other); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01NR014782-01A1 (NIH)
Record Dates: First submitted 2014-10-17; First posted 2014-11-06 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2014-10

CONDITIONS: HIV Health Literacy
Keywords: HIV/AIDS and HIV Testing Knowledge
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- English HIGH Health Literacy (Active Comparator): Using a valid measure of health literacy, 300 participants will be randomized into this group. These participants will receive HIV/AIDS and HIV testing information either by video or pictorial brochure in two equal groups.
  Interventions: Other: Video or Pictorial Brochure
- English LOW Health Literacy (Active Comparator): Using a valid measure of health literacy, 300 participants will be randomized into this group. These participants will receive HIV/AIDS and HIV testing information either by video or pictorial brochure in two equal groups.
  Interventions: Other: Video or Pictorial Brochure
- Spanish HIGH Health Literacy (Active Comparator): Using a valid measure of health literacy, 300 participants will be randomized into this group. These participants will receive HIV/AIDS and HIV testing information either by video or pictorial brochure in two equal groups.
  Interventions: Other: Video or Pictorial Brochure
- Spanish LOW Health Literacy (Active Comparator): Using a valid measure of health literacy, 300 participants will be randomized into this group. These participants will receive HIV/AIDS and HIV testing information either by video or pictorial brochure in two equal groups.
  Interventions: Other: Video or Pictorial Brochure

INTERVENTIONS:
Other: Video or Pictorial Brochure — Participants will receive HIV/AIDS and HIV testing information by video or by pictorial brochure according to patient health literacy level (lower or higher) and language (English or Spanish).

SUMMARY:
The Centers for Disease Control and Prevention (CDC) recommends that all patients should receive information about HIV/AIDS and HIV testing orally or in writing at every HIV testing encounter. However, for busy emergency departments (EDs), delivering information orally is a barrier to HIV testing, and written brochures likely are not useful for those with lower health or general literacy. Videos might be as or more efficacious than orally-delivered information in improving HIV/AIDS and HIV testing knowledge, particularly for those with lower health literacy skills. However, the resources required to show videos might limit their use in EDs. Pictorial brochures are a promising alternative, but are of unknown efficacy.

The objectives of this study are to: (1) determine if HIV/AIDS and HIV testing information should be delivered by a video or pictorial brochure to emergency department (ED) patients to improve short-term (in the ED) knowledge about HIV/AIDS and HIV testing; (2) determine if longer-term retention (over 12 months) of HIV/AIDS and HIV testing knowledge is greater for those who watch a video or review a pictorial brochure; (3) determine if short-term improvement and longer-term retention in HIV/AIDS and HIV testing knowledge is better after watching a video or reviewing a pictorial brochure for those with lower health literacy, and if improvement and retention also varies by language spoken (English or Spanish); and (4) if willingness to be tested again in one year is greater for those who watch the video or review the pictorial brochure, and if this willingness also varies by health literacy level and language spoken.

DETAILED DESCRIPTION:
Regardless of how patients are informed, the investigators do not know how well or for how long HIV/AIDS and HIV testing knowledge is retained, if this information should be delivered according to patient needs and abilities, and if retention of this knowledge impacts future HIV testing behavior.

The investigators will conduct a multi-site, randomized, controlled, longitudinal trial among 600 English- and 600 Spanish-speaking 18-64-year-old ED patients to investigate these questions. Using a valid measure of health literacy, the investigators will stratify our sample within language by health literacy level (lower vs. higher). The investigators will randomly assign patients to receive HIV/AIDS and HIV testing information by video or pictorial brochure. At one year post-enrollment, the investigators will offer participants an opportunity to be tested again for HIV.

At each study site (Birmingham,Cincinnati, Los Angeles, and Providence), the investigators will recruit 300 patients for a total of 1200 patients. Participants will be randomly assigned to receive HIV/AIDS and HIV testing information from a comparable pictorial brochure or a video. Randomization will be stratified by health literacy level (lower vs. higher) and language (English or Spanish). Those who are study eligible will undergo verbal consent to conduct the pre- and post-information questionnaires and information delivery portions of the study (video or pictorial brochure). No patient identifiers will be collected during the screening process, pre- or post-information questionnaires, or the information delivery phase of the study. For those who agree to be in the next portion of the study, written consent to participate will be obtained. Written consent will be obtained at this juncture because HIV testing and follow-up is performed, and because patient identifiers are needed for the remainder of the study. Participants will complete the study instruments at enrollment and at 3, 6, 9, and 12 months follow-up. At the end of one year, they will be offered the opportunity to be retested for HIV.

As primary aims, the investigators will compare the efficacy of pictorial brochures and videos in improving short-term (in ED) HIV/AIDS and HIV testing knowledge and retaining this knowledge over 12 months. More specifically, the investigators will determine if and how short-term improvement and longer-term retention of knowledge interacts with information delivery mode (pictorial brochure or video), patient health literacy level (lower or higher) and language (English or Spanish).

As secondary aims, using the Information-Motivation-Behavioral Skills (IMB model as a heuristic framework, the investigators will examine components of the IMB model relevant to our study and their interrelationships, their impact on HIV re-testing behavior, and the moderating influence of information delivery mode, language and health literacy level through the model. In regards to HIV re-testing behaviors, the investigators will assess: (1) testing uptake at one year post-enrollment when offered as part of the study, (2) testing utilization during the study period but not as part of the study, and (3) change in testing utilization one year pre vs. post study enrollment.

Study findings will guide ED-based delivery of HIV/AIDS and HIV testing information; that is, whether delivery modes (video or pictorial brochure) should be selected for patients by language and/or health literacy level, or whether either mode could be used. The results also will inform EDs when, how, and for whom information needs to be provided for those testing again for HIV within one year.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old; English or Spanish speaking

Exclusion Criteria:

* HIV positive; In an HIV vaccine trial; On HIV pre-exposure prophylaxis medication; In an HIV testing study; No personal telephone; Outside of the United States over next year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in HIV/AIDS and HIV testing knowledge questionnaire | Day 1
  The investigators will determine how short-term improvement of HIV/AIDS and HIV testing knowledge varies by information delivery mode (pictorial brochure or video), language (English or Spanish) and health literacy level (lower or higher) per four alternative hypotheses.
  Improvement of knowledge is:
  1. Greatest in the video arm who primarily speak English and have higher health literacy
  2. Greatest in the video arm among English speakers or higher health literacy patients
  3. Greater in the video arm than the pictorial brochure regardless of language and health literacy level
  4. The same despite information delivery mode, language, and health literacy level

SECONDARY OUTCOMES:
Change from Baseline in HIV/AIDS and HIV testing knowledge questionnaire at 12 months | 12 Months
  The investigators will determine how longer-term retention of HIV/AIDS and HIV testing knowledge varies by information delivery mode (pictorial brochure or video), language (English or Spanish) and health literacy level (lower or higher) per four alternative hypotheses.
  Retention of knowledge is:
  1. Greatest in the video arm who primarily speak English and have higher health literacy
  2. Greatest in the video arm among English speakers or higher health literacy patients
  3. Greater in the video arm than the pictorial brochure regardless of language and health literacy level
  4. The same despite information delivery mode, language, and health literacy level

CONTACTS AND LOCATIONS:
Overall Officials: Roland C Merchant, MD, Principal Investigator — Rhode Island Hospital

REFERENCES:
- [Derived] Merchant RC, Marks SJ, Clark MA, Carey MP, Liu T. Limited Ability of Three Health Literacy Screening Items to Identify Adult English- and Spanish-Speaking Emergency Department Patients With Lower Health Literacy. Ann Emerg Med. 2020 Jun;75(6):691-703. doi: 10.1016/j.annemergmed.2020.01.019. Epub 2020 Mar 20. PMID 32200999
- [Derived] Merchant RC, Liu T, Clark MA, Carey MP. Facilitating HIV/AIDS and HIV testing literacy for emergency department patients: a randomized, controlled, trial. BMC Emerg Med. 2018 Jul 9;18(1):21. doi: 10.1186/s12873-018-0172-7. PMID 29986662